CLINICAL TRIAL: NCT06848452
Title: Clinical Study on the Efficacy and Safety of Hydromorphone for ICU Analgesia
Status: Not yet recruiting | Type: Observational
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Other Study IDs: NTFY-YXY-01
Record Dates: First submitted 2025-02-14; First posted 2025-02-27 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Analgesia; ICU Patients Requiring Invasive Mechanical Ventilation
Keywords: ICU; hydromorphone; analgesia; remifentanil; sedation; respirator support
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients treated with hydromorphone and midazolam
  Interventions: Other: no-intervention
- Patients treated with remifentanil and midazolam
  Interventions: Other: no-intervention

INTERVENTIONS:
Other: no-intervention — no-intervention

SUMMARY:
This study is a prospective, single-center clinical study to evaluate the advantages, extensibility and safety of hydromorphone as an analgesic drug in ICU, and to compare it with remifentanil, a traditional sedative drug. These conclusions can guide us to understand the characteristics of analgesic drugs, carry out appropriate pain management, improve the status of ICU patients, and improve the quality of life of patients.

DETAILED DESCRIPTION:
This study will be carried out in the Affiliated Hospital of Nantong University. It is expected that 300 ICU patients who received invasive mechanical ventilation and needed analgesia and sedation will be included. The RASS and CPOT scores of 300 patients after using hydromorphone or remifentanil were collected and stored in the clinical trial sample database to evaluate and record the relevant indicators of the subjects. The relevant medical records in clinical treatment were analyzed and studied. Each subject will be numbered and a separate medical record established.

The purpose of this prospective single-center observational clinical study is to : 1 ) evaluate the advantages, extensibility and safety of hydromorphone as an ICU analgesic ; 2 ) Compared with the traditional sedative drug remifentanil. Including gastrointestinal dysfunction, respiratory depression, sedative use, mechanical ventilation time, ICU hospitalization time, extubation failure rate, etc.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤75 years;
* For patients requiring sedation and analgesia in ICU, invasive mechanical ventilation time is expected to be ≥24 hours;
* Obtain informed consent from patients or family members.

Exclusion Criteria:

* Under 18 years of age, or over 75 years of age;
* pregnancy or breastfeeding;
* Known or suspected allergy to opioids (e.g., fentanyl, remifentanil, hydromorphone), butorphanol, midazolam.
* General anesthesia surgery within 48 hours;
* Acute bronchial asthma.
* Acute intestinal obstruction.
* General anesthesia surgery within 48 hours;
* ECG QT interval: male >450 mm seconds, female >470 ms.
* Failure to obtain informed consent or authorization;
* Participate in other exploratory clinical trials within 6 months prior to screening;
* Severe hemodynamic instability (requires epinephrine greater than 0.5ug/kg/min to maintain MAP>65mmHg, or malignant arrhythmias frequently occur)
* Use of monoamine oxidase inhibitors.
* Chronic pain requires long-term analgesics (>3 months).
* Severe, pre-existing substantial liver disease with clinically significant portal hypertension, Child-Pugh grade C cirrhosis, or acute liver failure;
* Patients with acute and chronic renal insufficiency requiring dialysis treatment;
* Severe craniocerebral injury, brain tumor, increased intracranial pressure, cerebrovascular accident, coma, epileptic status, etc.
* Patients with a history of alcohol or drug abuse;
* Any condition that prevents the correct assessment of cognitive function, such as speech and sensory disorders or mental disorders (language difficulties or organic mental dysfunction);
* any other conditions which the investigator considers inappropriate for registration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients undergoing invasive mechanical ventilation requiring analgesia and sedation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
RASS score | The RASS score at 5, 10, 30 minutes and 1, 2, 3, 4, 8, 12, 16, 20, 24 hours post- dose and before and after each dose adjustment.
  Richmond Agitation and Sedation Scale score was used to assess the patient's calm state.The maximum value of the score table is 5 and the minimum value is - 4， indicating that the patient 's sedation level changes from ' coma ' to ' aggressive '.The higher the score, the worse the patient 's sedation depth and sedation quality.
CPOT score | The CPOT score at 5, 10, 30 minutes and 1, 2, 3, 4, 8, 12, 16, 20, 24 hours post- dose and before and after each dose adjustment.
  Critical care Pain Observation Tool score is used to evaluate the degree of pain in critically ill patients.The maximum value of the score table is 10, and the minimum value is 0.The higher the score, the more serious the pain of the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Department of Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Researchers hope to study data confidentiality.

REFERENCES:
- [Background] Muellejans B, Lopez A, Cross MH, Bonome C, Morrison L, Kirkham AJ. Remifentanil versus fentanyl for analgesia based sedation to provide patient comfort in the intensive care unit: a randomized, double-blind controlled trial [ISRCTN43755713]. Crit Care. 2004 Feb;8(1):R1-R11. doi: 10.1186/cc2398. Epub 2003 Nov 20. PMID 14975049
- [Background] Telekes A. [The role of hydromorphone in pain killing]. Lege Artis Med. 2008 Oct;18(10):675-9. Hungarian. PMID 19227610
- [Background] Hagen N, Thirlwell MP, Dhaliwal HS, Babul N, Harsanyi Z, Darke AC. Steady-state pharmacokinetics of hydromorphone and hydromorphone-3-glucuronide in cancer patients after immediate and controlled-release hydromorphone. J Clin Pharmacol. 1995 Jan;35(1):37-44. doi: 10.1002/j.1552-4604.1995.tb04743.x. PMID 7538514
- [Background] Inturrisi CE. Clinical pharmacology of opioids for pain. Clin J Pain. 2002 Jul-Aug;18(4 Suppl):S3-13. doi: 10.1097/00002508-200207001-00002. PMID 12479250
- [Background] Christrup LL. Morphine metabolites. Acta Anaesthesiol Scand. 1997 Jan;41(1 Pt 2):116-22. doi: 10.1111/j.1399-6576.1997.tb04625.x. PMID 9061094
- [Background] Panzer O, Moitra V, Sladen RN. Pharmacology of sedative-analgesic agents: dexmedetomidine, remifentanil, ketamine, volatile anesthetics, and the role of peripheral mu antagonists. Crit Care Clin. 2009 Jul;25(3):451-69, vii. doi: 10.1016/j.ccc.2009.04.004. PMID 19576524
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Lombardi RA, Pereira EM, Amaral S, Medeiros HJS, Alrayashi W. Erector spinae plane block versus intravenous opioid for analgesia in pediatric cardiac surgery: A systematic review and meta-analysis. Paediatr Anaesth. 2025 Jan;35(1):17-24. doi: 10.1111/pan.15027. Epub 2024 Oct 15. PMID 39403896
- [Background] Rahu MA, Grap MJ, Ferguson P, Joseph P, Sherman S, Elswick RK Jr. Validity and sensitivity of 6 pain scales in critically ill, intubated adults. Am J Crit Care. 2015 Nov;24(6):514-23. doi: 10.4037/ajcc2015832. PMID 26523009
- [Background] Hinkelbein J, Lamperti M, Akeson J, Santos J, Costa J, De Robertis E, Longrois D, Novak-Jankovic V, Petrini F, Struys MMRF, Veyckemans F, Fuchs-Buder T, Fitzgerald R. European Society of Anaesthesiology and European Board of Anaesthesiology guidelines for procedural sedation and analgesia in adults. Eur J Anaesthesiol. 2018 Jan;35(1):6-24. doi: 10.1097/EJA.0000000000000683. PMID 28877145
- [Background] Bauerschmidt A, Al-Bermani T, Ali S, Bass B, Dorilio J, Rosenberg J, Al-Mufti F. Modern Sedation and Analgesia Strategies in Neurocritical Care. Curr Neurol Neurosci Rep. 2023 Apr;23(4):149-158. doi: 10.1007/s11910-023-01261-7. Epub 2023 Mar 7. PMID 36881257
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131